CLINICAL TRIAL: NCT03285568
Title: Patterns of Prescribing and Monitoring of Palbociclib
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16082509
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Breast Cancer; Advanced Breast Cancer; Estrogen Receptor-positive Breast Cancer; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Palbociclib: women at least 18 years old, with ER+, HER2- advanced breast cancer, and were receiving palbociclib
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — Observe patients receiving palbociclib for dose adjustment and lab monitoring
  Other Names: IBRANCE

SUMMARY:
The purpose of this study is to determine if patients with ER+, human epidermal growth factor 2 negative (HER2-), advanced breast cancer are receiving dosing adjustments and monitoring based on manufacturer recommendations at a tertiary academic medical center.

DETAILED DESCRIPTION:
This study was a retrospective, single-center study that included women receiving palbociclib for the treatment of ER+, HER2- advanced breast cancer. Exclusion criteria were the presence of brain metastases or active enrollment in a palbociclib clinical trial.

The primary endpoint was the proportion of patients who were maintained on a palbociclib dose according to the adjustment schedule in package insert recommendations.

The secondary endpoints were the number of patients dose adjusted for hematologic toxicities, the number of patients experiencing neutropenia, duration of therapy, progression-free survival (PFS), and adherence to manufacturer monitoring recommendations.

ELIGIBILITY:
Inclusion Criteria:

* women at least 18 years old
* ER+, HER2- advanced breast cancer
* receiving palbociclib

Exclusion Criteria:

* brain metastases
* on palbociclib clinical trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women at least 18 years old with - ER+, HER2- advanced breast cancer
Study Population: All patients seen at RUMC
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Palbociclib dose according to the package insert recommendations. | 22 months
  Identify the proportion of patients who were maintained on a palbociclib dose according to the package insert recommendations.

SECONDARY OUTCOMES:
Dose adjustment for hematologic toxicities | 22 months
  Number of patients who required dose adjustment for hematologic toxicities while on the study.
Number of patients who experienced neutropenia. | 22 months
  Patients who experienced neutropenia as a result of their participation in the study.
Duration of therapy | 22 months
  Number of patients who completed the study compared to the number of patients who were was discontinued with the most common reason for discontinuation being disease progression
Progression free survival (PFS) | 22 months
  Progression free survival duration of patients that were in the study who received Palbociclib
Adherence to manufacturer monitoring recommendations | 22 months
  Patient adherence was also a limitation of this study as providers relied on the patient report to track medication adherence. Insurance coverage and access to palbociclib also contributed some variability as there were occasional delays in initiation of therapy or change in dose.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schultz, Principal Investigator — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: No